CLINICAL TRIAL: NCT00844701
Title: Validation of Cue Induced Imaging Paradigm in Nicotine Dependent Smokers
Brief Title: Cue Induced Imaging in Nicotine Dependent Smokers
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Karen Hartwell, M.D., Medical University of South Carolina - Clinical Neuroscience Division
Other Study IDs: BOLD fMRI
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2009-10

CONDITIONS: Nicotine Dependence
Keywords: nicotine; addiction; fMRI; neuroimaging; neurobiology; craving
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-smoker: Non-smoking control
- Nicotine Dependent Smoking Group: current smokers

SUMMARY:
The purpose of this study is to evaluate the relationship between craving to smoke and areas activated in brain. The researchers are using functional magnetic resonance imaging (MRI) that measures brain blood flow, or perfusion, to study this brain activation.

DETAILED DESCRIPTION:
Functional magnetic resonance imaging has demonstrated that the same types of environmental cues that induce craving activate an integrated network of brain areas involved in the appetitive and motivational process of addiction to drugs of abuse including nicotine ( Brieter 119; Koob 2001, Volkow 2003).In nicotine deprived smokers both mesolimbic dopamine reward pathways (amygdala, ventral tegmental area, and medial thalamus) and areas related to visuospatial attention (bilateral prefrontal cortex and parietal cortex and right fusiform gyrus) are activated by exposure to smoking images (Due 2002, David 2005).

In line with the National Institute on Drug Abuse's (NIDA) emphasis on novel methods for investigating substance use disorders, the current study proposes to use fMRI to better understand the neurological correlates of cue reactivity among nicotine dependent smokers. This approach will permit the isolation of pathways that are relevant to cue induced craving.

ELIGIBILITY:
Inclusion Criteria (nicotine dependent smoking group):

1. Age 18 - 60.
2. Participants will meet criteria for primary nicotine dependence, smoke at least 70% of days in the last 30 days prior to assessment.
3. Able to read and understand questionnaires and informed consent.
4. Right-handed.
5. Currently is not engaged in, and does not want, treatment for nicotine related problems.
6. Able to maintain abstinence from nicotine during the study period.
7. Participants must have a negative rapid-screening UDS and pregnancy test prior to imaging session.

Inclusion Criteria (nonsmoking control group):

1. Age 18 - 60.
2. Does not meet the DSM-IV criterion for lifetime or current substance dependence.
3. Has used tobacco products no more than on experimental basis (none in past year).
4. Participants must have a negative rapid-screening UDS and pregnancy test prior to session.
5. Righthanded.

Exclusion Criteria (all participants):

1. Currently meets DSM-IV criteria for any other psychoactive substance dependence disorder except nicotine dependence.
2. Any psychoactive substance abuse within the last 30 days as evidenced by subject report or urine drug screen.
3. Meets DSM-IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post-traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder. The rationale for excluding them is that symptoms from these disorders may affect dependent variables and complicate interpretation of the data.
4. Has current suicidal ideation with plan or homicidal ideation.
5. Need for maintenance or acute treatment with any psychoactive medication including antiseizure medications.
6. Clinically significant medical problems such as cardiovascular, renal, GI, or endocrine problem that would impair participation or limit ability to participate in scan.
7. Sexually active females of child-bearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
8. Has current charges pending for a violent crime (not including DUI related offenses).
9. Persons with ferrous metal implants or pacemaker since fMRI will be used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult nicotine dependent smokers
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hartwell, MD, Principal Investigator — Medical Universtiy of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States